CLINICAL TRIAL: NCT04537728
Title: My Healthy Brain: Preserving and Promoting Brain Health Through Evidence-based Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Ana-Maria Vranceanu, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019P003657
Record Dates: First submitted 2020-08-18; First posted 2020-09-03 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Aging; Mild Cognitive Impairment; Dementia; Old Age; Dementia; Cognitive Decline
Keywords: health; behavioral medicine; clinical psychology
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- My Healthy Brain Version 2 (Experimental): an 8-week group program that directly targets multiple lifestyle factors associated with brain health and prevention of CD
  Interventions: Behavioral: My Healthy Brain Version 2

INTERVENTIONS:
Behavioral: My Healthy Brain Version 2 — multimodal lifestyle intervention incorporating mindfulness skills, behavioral principles, and recent research on brain disease risk factors
  Other Names: MHBv2

SUMMARY:
The objective of this trial is to demonstrate early proof-of-concept for My Healthy Brain, an 8-week group program that directly targets multiple lifestyle factors associated with brain health and prevention of cognitive decline. The investigators will explore the feasibility, acceptability, and effect sizes of improvement in primary lifestyle outcomes as well as secondary outcomes of self-determination and subjective well-being.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* English fluency/literacy
* ≥1 modifiable brain disease risk factor (outlined by JAMA)
* Bluetooth 4.0 enabled smartphone

Exclusion Criteria:

* Diagnosis of dementia; Montreal Cognitive Assessment < 18
* Serious medical illness expected to worsen in next 6 months
* Current suicidal ideation
* Substance abuse
* Untreated serious mental health conditions
* Current use of digital monitoring device (eg. Fitbit)
* Mindfulness practice (> 45 minutes/week) in the last three months

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Credibility and Expectancy Questionnaire (CEQ) | Baseline (0 Weeks)
  percent of participants that score beyond scale midpoint
Client Satisfaction Questionnaire (CSQ-3) | Baseline (0 Weeks), Post-Test (8 Weeks)
  Items are summed to generate a total score; scores range from 3 to 12, with higher values indicating higher satisfaction.
Recruitment Feasibility | Baseline (0 Weeks)
  percent of referred patients meeting criteria to participate
Program Acceptability | Baseline (0 Weeks), Post-Test (8 Weeks)
  percent of participants completing at least 6 sessions
Treatment Fidelity | Baseline (0 Weeks), Post-Test (8 Weeks)
  percent of sessions rated as 100% adherent
Assessment Feasibility | Baseline (0 Weeks), Post-Test (8 Weeks)
  percent of post-questionnaires completed
Adherence to Actigraph | Baseline (0 Weeks), Post-Test (8 Weeks)
  percent of participants wearing Actiwatch ≥ 5 days per week
Adherence to Lifestyle Behaviors | Baseline (0 Weeks), Post-Test (8 Weeks)
  percent of participants completing weekly homework

SECONDARY OUTCOMES:
Change in Healthy Aging | Baseline (0 Weeks), Post-Test (8 Weeks)
  change from baseline to post test; measured by Brain Health Behaviors Checklist
Mindfulness: Cognitive and Affective Mindfulness Scale | Baseline (0 Weeks), Post-Test (8 Weeks)
  change from baseline to post test; Scores range from 12-48, with higher values reflecting greater mindfulness qualities.
Mindfulness: Homework log | Baseline (0 Weeks), Post-Test (8 Weeks)
  change from baseline to post test; measured by self-reported number of minutes practiced
Mindfulness: Five-Facet Mindfulness Questionnaire | Baseline (0 Weeks), Post-Test (8 Weeks)
  change from baseline to post test; Scores range from 15-75, with higher scores indicating greater mindfulness.
Sleep: Pittsburgh Sleep Quality Index | Baseline (0 Weeks), Post-Test (8 Weeks)
  change from baseline to post test;Total scores range from 0 to 21, with higher scores indicating greater sleep disturbance.
Sleep: Jenkins Sleep Questionnaire | Baseline (0 Weeks), Post-Test (8 Weeks)
  change from baseline to post test; scores range from 0-20, with higher scores indicating greater sleep disruption.
Sleep: Actigraph measures of sleep | Baseline (0 Weeks), Post-Test (8 Weeks)
  change from baseline to post test
Physical Activity: PROMIS Physical Function | Baseline (0 Weeks), Post-Test (8 Weeks)
  change from baseline to post test; scores range from 4-16, with higher scores signifying greater physical function.
Physical Activity: Godin Leisure Time Exercise Questionnaire | Baseline (0 Weeks), Post-Test (8 Weeks)
  change from baseline to post test; scores range from 0 to no upper limit, with higher scores indicating greater activity level.
Physical Activity: Rapid Assessment of Physical Activity | Baseline (0 Weeks), Post-Test (8 Weeks)
  change from baseline to post test; the highest score with an affirmative response is used for scoring, with higher scores indicating greater physical activity.
Physical Activity: Actigraph measures of activity | Baseline (0 Weeks), Post-Test (8 Weeks)
  change from baseline to post test
Nutrition: Mediterranean Eating Pattern for Americans Screener | Baseline (0 Weeks), Post-Test (8 Weeks)
  change from baseline to post test; scores range from 0-16, with higher scores indicating a greater adherence to the Mediterranean diet.
Nutrition: MIND Diet Adherence Checklist | Baseline (0 Weeks), Post-Test (8 Weeks)
  change from baseline to post test; scores range greater than or equal to 0, with higher scores indicating creater adherence to MIND diet.
Medication and Substance Use: Morisky Medication Adherence Scale | Baseline (0 Weeks), Post-Test (8 Weeks)
  change from baseline to post test; scores range from 0-4 with higher scores indicating greater adherence to medication regiment.
Medication and Substance Use: Alcohol Use Disorders Identification Test-Consumption | Baseline (0 Weeks), Post-Test (8 Weeks)
  change from baseline to post test; Scores range from 0-12, with higher scores indicating more hazardous drinking.
Medication and Substance Use: Fagerstrom Test for Nicotine Depedence | Baseline (0 Weeks), Post-Test (8 Weeks)
  change from baseline to post test; scores range from 0-10, with higher total scores indicating greater physical dependence on nicotine.
Stress and Emotional Functioning: Perceived Stress Scale | Baseline (0 Weeks), Post-Test (8 Weeks)
  change from baseline to post test; scores range from 0-40, with higher scores indicating greater perceived stress.
Stress and Emotional Functioning: PROMIS Depression | Baseline (0 Weeks), Post-Test (8 Weeks)
  change from baseline to post test; scores range from 8-40, with higher scores indicating greater depression.
Stress and Emotional Functioning: PROMIS Anxiety | Baseline (0 Weeks), Post-Test (8 Weeks)
  change from baseline to post test; scores range from 8-40, with higher scores indicating greater anxiety.
Stress and Emotional Functioning: Heart Rate Variability (Actigraphy) | Baseline (0 Weeks), Post-Test (8 Weeks)
  change from baseline to post test
Social Functioning: PROMIS Social Isolation | Baseline (0 Weeks), Post-Test (8 Weeks)
  change from baseline to post test; scores range from 6-30, with higher scores indicating greater social isolation.
Social Functioning: PROMIS Emotional Support | Baseline (0 Weeks), Post-Test (8 Weeks)
  change from baseline to post test; scores range from 4-16, with higher scores indicating lower emotional support.
Social Functioning: UCLA Loneliness Scale | Baseline (0 Weeks), Post-Test (8 Weeks)
  change from baseline to post test; scores range from 0-24, with higher scores indicating stronger perceptions of loneliness and social isolation.
Cognitive Functioning: Everyday Cognition Scale | Baseline (0 Weeks), Post-Test (8 Weeks)
  change from baseline to post test; scores range from 12-60, with higher scores indicating worse cognitive ability to perform everyday tasks.
Cognitive Functioning: PROMIS Cognition | Baseline (0 Weeks), Post-Test (8 Weeks)
  change from baseline to post test; scores range from 8-40, with higher scores indicating greater patient-perceived cognitive deficits.
Cognitive Functioning: Montreal Cognitive Assessment | Baseline (0 Weeks), Post-Test (8 Weeks)
  change from baseline to post test; scores range from 0-30, with higher scores representing greater global cognitive capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Maria Vranceanu, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schroeder MW, Frumkin MR, Mace RA. Proof-of-concept for integrating multimodal digital health assessments into lifestyle interventions for older adults with dementia risk factors. J Behav Med. 2025 Apr;48(2):373-384. doi: 10.1007/s10865-024-00546-7. Epub 2025 Jan 20. PMID 39833389